CLINICAL TRIAL: NCT03852927
Title: Computer Guided Contouring of Craniofacial Fibrous Dysplasia Involving Zygoma: a Case Series
Brief Title: Computer Guided Contouring of Craniofacial Fibrous Dysplasia Involving Zygoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sherif Ali, Lecturer of oral and maxillofacial surgery, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-1-20
Record Dates: First submitted 2019-02-22; First posted 2019-02-25 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Craniofacial Fibrous Dysplasia
MeSH Terms: conditions — Craniofacial Fibrous Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Computer guided contouring — Using virtual planing and rapid prototyping a surgical guide will be fabricated, and will be used for bone contouring of the bone lesion.
  Other Names: Computer guided shaving

SUMMARY:
This study will be conducted on patients with monostotic unilateral craniofacial fibrous dysplasia affecting zone I (fronto-orbital, zygomatic, and upper maxillary regions). Computer guided shaving will be performed for all the patients, and the accuracy of this procedure will be assessed.

DETAILED DESCRIPTION:
This study will be conducted on patients with monostotic unilateral craniofacial fibrous dysplasia affecting zone I (fronto-orbital, zygomatic, and upper maxillary regions).

I. Preoperative preparation

1. Virtual planning Computed tomography (CT) will be performed for the skull using a multi-slice helical CT machine. Computed tomography DICOM (digital Imaging and Communication in Medicine) files will be imported to the 3D surgical planning software (Mimics 10.0, Materialise NV, Leuven, Belgium). Using the software and through a series of segmentation and simulation processes, area of interest will be virtually selected and separated. Finally, the virtual image of the surgical guide will be reconstructed.
2. Rapid prototyping Stereolithographic (STL) files of the virtual image will be exported to multi-jet modelling printing machine (InVision Si2, 3D Systems e Rock Hill, SC) and will be fabricated using plastic material (VisiJet SR 200, 3D Systems e Rock Hill, SC).

II. Surgical procedures Area of interest for all patients will be exposed using the hemicoronal, and maxillary intraoral vestibular incisions. The surgical guide(s) will be seated in position on the affected side. Bone removal will be performed through the guide according to the preoperative planning. The bone removal will be then performed to connect the guiding holes using surgical burs. Finally, the incisions will be sutured after soft tissue suspension.

III. Follow up Postoperative CT will be performed for postoperative assessment. After 1 week patients will be recalled for suture removal and clinical assessment. Then the patients will be recalled 1, 3 months for further assessment.

ELIGIBILITY:
Inclusion Criteria:

* Monostotic unilateral craniofacial fibrous dysplasia.
* Facial asymmetry affecting zone I (fronto-orbital, zygomatic, and upper maxillary regions)
* More than 17 years

Exclusion Criteria:

* functional deficits
* orbital manifestations

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2019-01-25 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Accuracy | 1 week after the surgical procedure
  Preoperative plane and post-operative 3D CT scan will superimposed, and the difference between the planed and postoperative bone contour will be estimated.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry, Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided